CLINICAL TRIAL: NCT04010032
Title: The Effect of Programmed Intermittent Epidural Bolus Versus Continuous Epidural Infusion on Postoperative Analgesia in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 4-2019-0418
Record Dates: First submitted 2019-06-25; First posted 2019-07-08 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Correctional Osteotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: triple (Participant, Care Provider, investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIEB (Programmed intermittent epidural bolus) (Experimental): bolus administration of 0.15 ml of ropivacaine 0.15 ml / kg into epidural space every hour(intermittent bolus injection)
  Interventions: Device: Programmed intermittent epidural bolus
- CEI (Continuous epidural infusion) (Active Comparator): Continuous infusion of 0.15% ropivacaine 0.15 ml / kg / h into the epidural space using PCA device
  Interventions: Device: Continuous epidural infusion

INTERVENTIONS:
Device: Programmed intermittent epidural bolus — bolus administration of 0.15 ml of ropivacaine 0.15 ml / kg into epidural space every hour(intermittent bolus injection) using PCA device
  Other Names: PIEB
  Arms: PIEB (Programmed intermittent epidural bolus)
Device: Continuous epidural infusion — Continuous infusion of 0.15% ropivacaine 0.15 ml / kg / h into the epidural space using PCA device using PCA device
  Other Names: standard, CEI
  Arms: CEI (Continuous epidural infusion)

SUMMARY:
The aim of this study was to compare the efficacy of a programmed intermittent bolus injection method compared to conventional continuous infusion in the management of epidural analgesia in pediatric patients correctional osteotomy. As a prospective double blinded randomized controlled trial, the investigators compare the quality of pain control after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pediatric patients with between 4 and 13 years
* 2. Patients scheduled for correctional osteotomy of the lower extremity
* 3. Pediatric patients whose weight of 40kg of less

Exclusion Criteria:

* 1. Contraindications to epidural analgesia (local infection, blood clotting disorder, anatomical abnormality, sepsis, etc.)
* 2. Patients with symptoms/signs of elevated intracranial pressure with or without a history of elevated intracranial pressure
* 3. If all of the parents of the subject are foreigners or illiterate (if the parents of the subject can not read the agreement)

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Difference in total amount of ropivacaine injected through epidural analgesia | 6 hours after surgery
  The difference in the amount of ropivacaine injected into epidural space for 6 hours postoperatively
Difference in total amount of ropivacaine injected through epidural analgesia | 12 hours after surgery
  The difference in the amount of ropivacaine injected into epidural space for 12 hours postoperatively
Difference in total amount of ropivacaine injected through epidural analgesia | 24 hours after surgery
  The difference in the amount of ropivacaine injected into epidural space for 24 hours postoperatively
Difference in total amount of ropivacaine injected through epidural analgesia | 36 hours after surgery
  The difference in the amount of ropivacaine injected into epidural space for 36 hours postoperatively
Difference in total amount of ropivacaine injected through epidural analgesia | 48 hours after surgery
  The difference in the amount of ropivacaine injected into epidural space for 48 hours postoperatively

SECONDARY OUTCOMES:
The time for the first patient controlled rescue epidural bolus after surgery | 48 hours after surgery
Number of patient-controlled rescue epidural bolus for 48 hours postoperatively | 48 hours after surgery
Pain scores for 6 hours after surgery (VAS) | 6 hours after surgery
  VAS(visual analogue scale) :0(no paine)~10(wort possible, unbearable, excruciating apin)
Pain scores for 12 hours after surgery (VAS) | 12 hours after surgery
  VAS(visual analogue scale) :0(no paine)~10(wort possible, unbearable, excruciating apin)
Pain scores for 24 hours after surgery (VAS) | 24 hours after surgery
  VAS(visual analogue scale) :0(no paine)~10(wort possible, unbearable, excruciating apin)
Pain scores for 48 hours after surgery (VAS) | 48 hours after surgery
  VAS(visual analogue scale) :0(no paine)~10(wort possible, unbearable, excruciating apin)
Pain scores for 6 hours after surgery (r-FLACC) | 6 hours after surgery
  r-FLACC scale (revised Face, Legs, Activity, Cry, Consolability scale): summation of each items and total range is 0~10. higher values represent a more severe pain.
Pain scores for 12 hours after surgery (r-FLACC) | 12 hours after surgery
  r-FLACC scale (revised Face, Legs, Activity, Cry, Consolability scale): summation of each items and total range is 0~10. higher values represent a more severe pain.
Pain scores for 24 hours after surgery (r-FLACC) | 24 hours after surgery
  r-FLACC scale (revised Face, Legs, Activity, Cry, Consolability scale): summation of each items and total range is 0~10. higher values represent a more severe pain.
Pain scores for 48 hours after surgery (r-FLACC) | 48 hours after surgery
  r-FLACC scale (revised Face, Legs, Activity, Cry, Consolability scale): summation of each items and total range is 0~10. higher values represent a more severe pain.
Whether to administer additional intravenous narcotic analgesics with total additional intravenous analgesic dose. | 48 hours after surgery
  -% of patients with given intravenous additional narcotic analgesics
  * number of administrating intravenous additional narcotic analgesics per patient
Whether to administer additional intravenous narcotic analgesics with total additional intravenous analgesic dose. | 48 hours after surgery
  -% of patients with given intravenous additional narcotic analgesics
  * total additional dose of intravenous narcotic analgesics per patient
Whether to administer additional intravenous narcotic analgesics with total additional intravenous analgesic dose. | 48 hours after surgery
  -% of patients with given intravenous additional narcotic analgesics
  * measurement tool: Electronic Medical Record(including Drug administration history)
A dull feeling the patient feels | 6 hours after surgery
  A dull feeling the patient feels : yes or no
A dull feeling the patient feels | 12 hours after surgery
  A dull feeling the patient feels : yes or no
A dull feeling the patient feels | 24 hours after surgery
  A dull feeling the patient feels : yes or no
A dull feeling the patient feels | 48 hours after surgery
  A dull feeling the patient feels : yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No